CLINICAL TRIAL: NCT04221243
Title: Evaluation Of Innovative 3D Printed Space Maintainer Versus Conventional One
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Farah Ahmed Barakat (Other)
Responsible Party: Sponsor-Investigator, Farah Ahmed Barakat, Teaching Assistant in British University in Egypt, British University In Egypt
Organization: British University In Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PED-4M
Record Dates: First submitted 2019-10-01; First posted 2020-01-09 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Missing Teeth
Keywords: space maintainer; 3D printing
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Children with 3D printed space maintainer (Experimental)
  Interventions: Device: 3D printed space maintainer by NextDent Ortho Rigid
- Group 2: Children with conventional band and loop (Active Comparator)
  Interventions: Device: Conventional Band and Loop

INTERVENTIONS:
Device: 3D printed space maintainer by NextDent Ortho Rigid — Biocompatible 3D printing material
  Arms: Group 1: Children with 3D printed space maintainer
Device: Conventional Band and Loop — metal space maintainer
  Arms: Group 2: Children with conventional band and loop

SUMMARY:
The primary aim of this study is to introduce a new effective and efficient 3D printed design of an intra-oral space maintainer.

The secondary aim of the study is to:

Evaluate the clinical performance of 3D printed space maintainer versus conventional metal band and loop over a period of 6 months regarding their functional , biological aspects and patient satisfaction.

DETAILED DESCRIPTION:
And will be conducted as follows:

* In-Vivo evaluation of the clinical performance of 3D printed space maintainer versus metal band and loop concerning oral hygiene, retention and patient satisfaction.
* A total of thirty healthy subjects will be selected from the Pediatric Dentistry and Dental Public Health outpatient clinic, Faculty of Dentistry, Ain Shams University. They will be divided using simple randomization in two groups:

Group 1: Children with 3D printed space maintainer (n=15) Group 2: Children with conventional band and loop(n=15)

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-9years' old
* Premature loss of primary molar or molars in one or more quadrant.
* Absence of abnormal dental conditions such as cross bite.
* Sound and healthy buccal and lingual surfaces of abutment teeth.

Exclusion Criteria:

* Bad oral hygiene
* Medically Compromised patients.
* Presence of periapical pathology radiographically.
* Carious buccal and lingual surfaces of abutment teeth.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
introduce a new 3D printed design of an intraoral space maintainer. | 6 months
  The function of the new intraoral space maintainer will be assessed whether good retention is obtained or not,by checking whether it fell off the patient's mouth or not .

SECONDARY OUTCOMES:
compare between the new 3D printed space maintainer versus conventional metal band and loop regarding their biological aspects. | 6 months
  Biologically, the oral hygiene of the patient will be assessed by measuring the plaque and the gingival indices scores on the corresponding teeth on a scale from 0-3
compare between the new 3D printed space maintainer versus conventional metal band and loop regarding their patient satisfaction. | 6 months
  Patient satisfaction will be assessed by a satisfaction questionnaire given to the patient (scale from 1-3)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No